CLINICAL TRIAL: NCT03772483
Title: Efficacy of Virtual Reality Distraction in Reducing Injection Pain and Anxiety During Local Anesthesia in Pediatric Dental Patients
Brief Title: Efficacy of Virtual Reality in Reducing Injection Pain and Anxiety During Local Anesthesia in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Plovdiv Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PlovdivMU2
Record Dates: First submitted 2018-12-06; First posted 2018-12-11 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Injection Pain; Local Anesthesia
Keywords: virtual reality; pain control; pediatric dental patients; pediatric pain management; local anesthesia children
MeSH Terms: conditions — Agnosia | interventions — Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: Randomized Intervention Model: Split-mouth assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Local anesthesia with conventional syringe
  Interventions: Procedure: Local anesthesia with conventional syringe
- Virtual reality group (Active Comparator): Local anesthesia with conventional syringe + VR device
  Interventions: Device: Local anesthesia with conventional syringe + VR device

INTERVENTIONS:
Procedure: Local anesthesia with conventional syringe — Buccal infiltration in posterior maxillary region with traditional technique. A 27 gauge short needle is inserted in the mucobuccal fold above the tooth to be anesthetized.
  Local anesthetic infiltration speed 1ml/min. Drug: Local anaesthetic - Ubistesin - 4% Articaine with adrenaline 1: 200 000 1.7 mL
  Arms: Control group
Device: Local anesthesia with conventional syringe + VR device — Virtual reality device (Noon VR, Gear FX) is placed on the face of the patient, playing a video of soothing and peaceful natural landscapes.
  Buccal infiltration in posterior maxillary region with traditional technique. A 27 gauge short needle is inserted in the mucobuccal fold above the tooth to be anesthetized.
  Local anesthetic infiltration speed 1ml/min. Drug: Local anaesthetic - Ubistesin - 4% Articaine with adrenaline 1: 200 000 1.7 mL
  Arms: Virtual reality group

SUMMARY:
The aim of this study is to determine the efficacy of a virtual reality (VR) device in reducing injection pain and anxiety associated with local anesthesia in pediatric dental patients.

The clinical trial is a randomized split-mouth assignment. Included patients are 8-12 years old requiring local anesthetic infiltration with conventional syringe (CS) for conservative treatment of two primary maxillary molars bilaterally.

Eligible patients undergo two single-visit treatments after CFSS-DS measurement before each, whereas VR is allocated to either first or second local anesthesia procedure. Primary outcome measure will be pain felt during injection, reported by patient on visual analogue scale (VAS). Secondary outcome measures: self-reported anxiety during injection on FIS; pain-related behavior according to FLACC scale; heart-rate dynamics; patient preference to local anesthesia method - CS or CS+VR.

DETAILED DESCRIPTION:
Achieving local anesthesia in children is one of the critical aspects of pain management.

A contemporary engaging form of distraction is represented by virtual reality devices. Virtual reality (VR) devices create a virtual environment of view and sound that allow patients to be immersed in an interactive, simulated world to distract them from pain. The VR devices have a wide viewing field and three-dimensional displays that project the images right in front of the user. They not only show potentially attractive audio-visual stimuli, but also exclude all other visual environmental stimuli that may affect the patient.

The aim of this study is to determine the efficacy of a virtual reality (VR) device in reducing injection pain and anxiety associated with local anesthesia in pediatric dental patients.

The device used in this study is Noon VR, FXGear, compatible with a mobile phone.

The clinical trial is a randomized split-mouth assignment. Included patients are healthy positive children 8-12 years old requiring local anesthetic infiltration for conservative treatment of two primary maxillary molars bilaterally.

Eligible patients undergo two single-visit treatments after measurement of dental fear prior to each according to the Dental Subscale of the Children's Fear Survey Schedule (CFSS-DS). Local anesthetic is delivered through buccal infiltration with conventional syringe, where as the virtual reality distraction is allocated to either first or second local anesthesia procedure. Primary outcome measure will be pain felt during injection, reported by patient on visual analogue scale. Secondary outcome measures: self-reported anxiety during injection on Facial Image Scale; pain-related behavior according to Faces, Legs, Activity, Cry, Consolability (FLACC) scale; heart-rate dynamics; patient preference to local anesthesia method - traditional infiltration or virtual reality device-assisted injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients, identified as positive or definitely positive through Frankl behavioral rating scale.
* Children, requiring local anesthesia infiltration for conservative treatment of two primary upper jaw molars bilaterally.
* Children without previous experience with local anesthesia for dental treatment.
* Obtained informed consent from parents or gave-givers to participate in the study.

Exclusion Criteria:

* Children who are considered medically compromised or medically complex patients. The absence of disease is confirmed by anamnestic interview with a parent or a care-giver of the child and excludes general acute or chronic disease, cognitive impairment, psychogenic non-epileptic events, sensitivity to flashing light or motion.
* Vision requiring correction with eyeglasses.
* Recent injury to the eyes or face that prevents comfortable use of VR hardware or software.
* Patients who are undergoing therapy with neurological, sedative, analgesic and/or anti-inflammatory drugs 7 days prior to treatment.
* Patients with allergy to local anesthetics of the amide group.
* Children, who are first time ever dental patients.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Pain felt during injection using visual analogue scale | Immediately after local anesthetic delivery
  Self-reported pain by the patient immediately after local anaesthesia infiltration using a VAS (visual analogue scale), containing a combination of Numeric Rating Scale (0-10, where 0 means no pain, 10 - worst possible pain) and Wong-Baker Faces Pain Scale, including pictures of facial expressions with correlating numbers of 0-10 (0 being 'no hurt' and 10 being 'hurts worst'). The combination allows children to pick a facial expression, that corresponds with their pain and see a number that matches it.

SECONDARY OUTCOMES:
Pain-related behavior evaluated on the Faces, Legs, Activity, Cry, Consolability Behavioral Pain Rating Scale | During local anesthesia procedure
  Evaluated by the outcomes assessor. The FLACC scale has five criteria - Faces, Legs, Activity, Cry, Consolability, which are each assigned a score of 0, 1 or 2. Total score of scale is summed in range 0 to 10, where: 0=relaxed and comfortable; 1-3=mild discomfort; 4-6=moderate pain; 7-10=severe pain.
Self-reported anxiety during injection evaluated on FIS | Immediately after local anesthetic delivery
  The Facial Image Scale (FIS) comprises a row of five faces from very unhappy (score 5) to very happy (score 1).
Heart rate dynamics of the patient | Start: in the waiting room, at least 5 minutes before local anaesthesia procedure. End: at least 5 minutes after treatment.
  Patient's left index finger is connected to a portable recording pulse oximeter for children.
Assessment of self-reported dental fear on CFSS-DS questionnaire | At least 5 minutes before local anesthesia
  Assessment will be performed prior to both visits.
Patient preference to local anesthesia method | One week after second procedure
  One week after the second dental visit, the patient is reached by a phone call and asked: "Which method do you prefer to put your tooth to sleep? With the virtual reality device or without it?"

CONTACTS AND LOCATIONS:
Overall Officials: Elitsa Veneva, DMD, Principal Investigator — Plovdiv Medical University
Locations (1):
- Department of Pediatric Dentistry, Faculty of Dental Medicine, Plovdiv, Bulgaria

IPD SHARING:
Plan to Share IPD: No